CLINICAL TRIAL: NCT04676217
Title: Position Related Changes in Macular Hole Morphology Before and After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1917
Record Dates: First submitted 2020-11-27; First posted 2020-12-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDP (Active Comparator): Face down positioning
  Interventions: Procedure: Postoperative positioning advice
- NSP (Experimental): No positioning named "non-supine positioning". Participants are to avoid recumbent positioning.
  Interventions: Procedure: Postoperative positioning advice

INTERVENTIONS:
Procedure: Postoperative positioning advice — The postoperative positioning advice until 3 am the same day.

SUMMARY:
Macular hole is a full thickness retinal defect in the very centre of the retina that gives the sharpest vision. The condition causes a substantial deterioration of visual acuity, and operative measures are necessary in order to close the defect and improve the visual function. A macular hole has varying degrees of retinal oedema surrounding the hole edges. The oedema is maintained by continuous of liquid into the tissue and effectively prevents spontaneous closure. For that reason it is essential for macular hole closure that the macula has minimal contact with intraocular fluid in the very early postoperative phase. This is why the treatment included a long-lasting intraocular gas tamponade and typically, one week of face-down positioning (FDP) after surgery.Our aim is to investigate the impact of diurnal, orthostatic, and gravitational variations on macular hole morphology before and after surgery. The participants will be examinated with optical coherence tomography 8-10 am, 1 pm, and 3 pm. Between 8 am and 1 pm ,the patient is encouraged to an upright position. After the 1 pm examination, the patient will be positioned flat on the side of the eye with macular hole until the 3 pm examination. The surgery will be performed before 10 am. Postoperatively a randomization to face down positioning or no positioning until 3 am. Optical coherence tomography images through gas tamponade is made at 3 am.

ELIGIBILITY:
Inclusion Criteria:

* Primary macular hole
* Able to sign informed consent
* Signed informed consent

Exclusion Criteria:

* Previous vitreoretinal surgery in the study eye
* Secondary macular holes caused by other conditions than vitreomacular traction
* Myopic macular hole, i.e. excessive myopia (more than -6 dioptres)
* Posttraumatic macular hole
* Macular holes secondary to retinal detachment or other retinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Macular hole mid diameter | 1 day
  Micrometer
Macular hole basal diameter | 1 day
  Micrometer
Macular hole mid area | 1 day
  Square micrometer
Central retinal thickness | 1 day
  Micrometer

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Department of Ophthalmology, Stavanger

IPD SHARING:
Plan to Share IPD: No